CLINICAL TRIAL: NCT05204654
Title: A Comparison of Class II Correction Using the Carriere Motion Appliance Versus an In-Office Sectional Appliance: Treatment Effects and Efficiency
Brief Title: Carriere Motion Appliance* Versus In-office Sectional Appliance
Acronym: CMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough subjects were recruited for the study.
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Alexandria Mary Newton, Orthodontic Resident, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005827
Record Dates: First submitted 2021-12-22; First posted 2022-01-24 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Angle Class 2 Malocclusion
Keywords: Carriere Motion Appliance; Angle Class 2 Malocclusion

STUDY DESIGN:
Intervention Model Description: Subjects participating in the study and will then be randomly assigned to one of two treatment interventions:
  1. Sagittal first approach using the CMA
  2. Sagittal first approach using an in-office fabricated custom appliance
  At the bonding appointment, the appliance will be bonded and AP correction will begin. Both treatment groups will have a button bonded to the mandibular first molars, and Essix retainers with 2 mm thickness will require to be worn at all times for mandibular anchorage during AP correction (only taken out to brush and eat). Both treatment groups will follow the CMA protocol for Class II correction, which consists of wearing Force 1 (1/4, 6 oz) Class II elastics for the first month of treatment, and Force 2 (3/16, 8 oz) Class II elastics for the remainder of Class II correction. Once Class II correction is complete, the appliance will be removed and a lateral cephalometric radiograph and digital model will be obtained
Who Masked: Outcomes Assessor
Masking Description: Lateral cephalometric radiographs and digital study models will be de-identified prior to landmarking and obtaining measurements. The appliances will not be present on the patient when these records are obtained and therefore, when taking measurements, the outcomes assessor will not know which intervention the subjects received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- In-office fabricated appliance (Experimental): A customized in-office fabricated appliance using the printed digital model of the subject will be used for AP correction. AP correction will be completed following CMA protocol (see model description)
  Interventions: Other: In-office fabricated appliance
- Carriere Motion Appliance (Active Comparator): The appropriate length appliance will be placed as directed in the CMA handbook on the maxillary first molar and canine. AP correction will be completed following CMA protocol (see model description)
  Interventions: Device: Carriere Motion Appliance

INTERVENTIONS:
Other: In-office fabricated appliance — A 0.022 Slot MBT™ second molar mini tube that has been modified to have a 2 mm length will be placed on the maxillary first molar and a 0.018 slot MBT™ maxillary canine bracket will be placed on the maxillary canine, with a 0.016x0.022 stainless-steel wire spanning from the maxillary first molar to the maxillary canine. A bayonet bend will be placed mesial to the molar tube. A curve will be bent into the wire, so that the wire is able to passively rest on the buccal surface of the maxillary canine. A stainless-steel closed coil will span the molar to canine and lay flush to the mesial portion of the molar tube and the distal portion of the canine bracket. The wire will be cinched mesial to the maxillary canine tie-wing and also 2-3 mm distal to the maxillary first molar to ensure that the molar can rotate during treatment, if needed. A stainless-steel tie will be used to secure the wire into the canine bracket. AP correction will be completed following CMA protocol
  Arms: In-office fabricated appliance
Device: Carriere Motion Appliance — A bar spanning from the maxillary first molar to canine with a ball and socket joint at the molar and a canine pad at the canine. A slight bend is present between the molar and canine bracket. The ball and socket is designed to allow the molar to rotate to -15 degrees along it's longitudinal axis. The appliance claims that it allows for Class II correction with minimal secondary tooth movements when used with mandibular anchorage.
  Other Names: CMA
  Arms: Carriere Motion Appliance

SUMMARY:
The "sagittal first" approach to Class II correction in orthodontic treatment involves correcting the antero-posterior (AP) relationship of the maxillary and mandibular dentition prior to the leveling and aligning phase of orthodontic treatment. The Carriere Motion Appliance (CMA) was made to provide sagittal correction prior to orthodontic treatment with minimal secondary tooth movements that are typically seen with Class II correction. The aim in this study is to explore the efficacy and efficiency of Class II molar correction in adolescent patients using the sagittal first approach with either a sectional, in-office fabricated appliance or the CMA, by measuring total treatment duration (in months) as well as comparing dental and skeletal measurements taken from lateral cephalometric radiographs obtained prior to Class II correction (T0) and immediately after removal of the appliance (T1). The investigators will also be comparing secondary molar and canine rotational movements after Class II correction by comparing digital dental casts obtained at T0 and T1.

DETAILED DESCRIPTION:
The investigators will be recruiting 12 to 17-year 11-month old patients with a Class II molar relationship,who are presenting for comprehensive orthodontic treatment at the Postgraduate orthodontic clinic at University at Buffalo School of Dental Medicine. Recruited subjects will be randomized into one of 2 groups. Both groups will be receiving a method of Class II correction using the Sagittal First approach, which means the Class II molar relationship will be corrected prior to the leveling and aligning phase of orthodontic treatment. Subjects will be treated using either the Carriere Motion Appliance (CMA), or a sectional appliance fabricated with materials that are commonly found in orthodontic practice. Both appliances will be used according to the CMA guidelines. After Class II correction and removal of appliance, and prior to the next stage of treatment, an additional digital scan of the mouth and a lateral cephalometric radiograph will be taken. Dental and skeletal measurements from initial cephalometric radiographs and models will be subtracted from the corresponding measurements taken on radiographs and models obtained after Class II correction, and comparisons will be made between the two treatment treatment groups. Efficiency will be determined by number of months until Class II molar and canine correction was obtained, and efficacy will be determined by the skeletal and dental measurements obtained.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Presenting for comprehensive orthodontic treatment at the Postgraduate orthodontic clinic at the University at Buffalo School of Dental Medicine
* Unilateral or bilateral ½-cusp to full-cusp Class II molar and canine relationship
* Growing Patients (~12-17y 11m)
* Subjects who do not require extractions as part of treatment mechanics
* Mild to moderate crowding

Exclusion Criteria:

* Patients in mixed dentition
* Any missing teeth up to and including permanent first molars
* Bilateral molar relationship of less than ½ cusp Class II prior to appliance cementation

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Covell, DDS, PhD, Study Chair — Orthodontics Department Chair, University at Buffalo School of Dental Medicine
Locations (1):
- University at Buffalo School of Dental Medicine, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Study terminated due to time restraint | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14.5 [14 to 15] | 14.5 [14 to 15] | 14.5 [14 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Treatment Time
Description: Months
Time Frame: From date of Class II correction appliance delivery to date of removal of Class II correction appliance after Class I molar and canine relationship has been established (approximately 120-180 days).
Population: Data were not collected, study was terminated due to time constraint and no data on participants was collected.
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Skeletal Changes
Description: Degrees, Millimeters
Time Frame: as for outcome 1
Population: Data were not collected, study was terminated due to time constraint and no data on participants was collected.
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Dental Changes
Description: Degrees, Millimeters
Time Frame: as for outcome 1
Population: Data were not collected, study was terminated due to time constraint and no data on participants was collected.
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Maxillary Canine and Maxillary First Molar Rotation
Description: Degrees
Time Frame: as for outcome 1
Population: Data were not collected, study was terminated due to time constraint and no data on participants was collected.
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Deaths and adverse events were not collected
Description: Deaths and adverse events were not collected
Arm/Group | In-office Fabricated Appliance | Carriere Motion Appliance
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT05204654/Prot_000.pdf